CLINICAL TRIAL: NCT05338333
Title: Clinical Performance Evaluation of Two Frequent Replacement Silicone Hydrogel Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLN705-C001
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Presbyopia
Keywords: Contact lenses; Multifocal
MeSH Terms: conditions — Presbyopia | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LID210464, then AOHG MF (Other): Lehfilcon A multifocal contact lenses (LID210464) worn in Period 1, with lotrafilcon B multifocal contact lenses (AOHG MF) worn in Period 2, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 30 days. CLEAR CARE® will be used for nightly contact lens cleaning and disinfecting.
  Interventions: Device: Lehfilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses; Device: CLEAR CARE®
- AOHG MF, then LID210464 (Other): Lotrafilcon B multifocal contact lenses (AOHG MF) worn in Period 1, with lehfilcon A multifocal contact lenses (LID210464) worn in Period 2, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 30 days. CLEAR CARE® will be used for nightly contact lens cleaning and disinfecting.
  Interventions: Device: Lehfilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses; Device: CLEAR CARE®

INTERVENTIONS:
Device: Lehfilcon A multifocal contact lenses — Investigational frequent replacement soft contact lens indicated for the optical correction of presbyopia
  Other Names: LID210464
Device: Lotrafilcon B multifocal contact lenses — Commercially available frequent replacement soft contact lens indicated for the optical correction of presbyopia
  Other Names: AOHG MF; AIR OPTIX® plus HydraGlyde® Multifocal (AOHG MF) contact lenses
Device: CLEAR CARE® — Hydrogen peroxide-based contact lens cleaning and disinfecting solution

SUMMARY:
The primary objective of this study is to demonstrate noninferiority in visual acuity at distance when wearing the test contact lenses (LID210464) compared to the control contact lenses (AOHG MF) after 30 days of wear.

DETAILED DESCRIPTION:
Subjects will be expected to attend 4 office visits and will be dispensed study contact lenses (test lenses and control lenses) for a 30-day duration of bilateral wear for each study lens type (total of approximately 60 days of contact lens wear).

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an informed consent form that has been approved by an Institutional Review Board.
* Willing and able to attend all study visits as required by the protocol.
* Willing to stop wearing habitual contact lenses for the duration of the study.
* Currently wearing daily disposable and biweekly/monthly replacement multifocal soft contact lenses in both eyes at least 5 days per week and at least 8 hours per day for at least 3 months. AOHG MF wearers may be included.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any eye infection, inflammation, abnormality, or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator.
* History of refractive surgery or planning to have refractive surgery during the study.
* Current or history of pathologically dry eye.
* Currently pregnant or lactating.
* Other protocol-specified exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Kindred Optics at Maitland Vision, Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Kannarr Eye Care LLC, Pittsburg, Kansas
  - The Eye Doctors, Inc., Eden Prairie, Minnesota
  - Complete Eye Care of Medina, Medina, Minnesota
  - ProCare Vision Centers, Inc., Granville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all enrolled participants, as treated (101). Note, one subject that was randomized to AOHG MF, then LID210464 was exposed to LID210464, then AOHG MF instead.
Units Other Than Participants: eyes
Groups:
- LID210464, Then AOHG MF: Lehfilcon A multifocal contact lenses (LID210464) worn in Period 1, with lotrafilcon B multifocal contact lenses (AOHG MF) worn in Period 2, as randomized. Each study lens type was worn bilaterally (in both eyes) for 30 days. CLEAR CARE® was used for daily contact lens cleaning and disinfecting.
- AOHG MF, Then LID210464: Lotrafilcon B multifocal contact lenses (AOHG MF) worn in Period 1, with lehfilcon A multifocal contact lenses (LID210464) worn in Period 2, as randomized. Each study lens type was worn bilaterally (in both eyes) for 30 days. CLEAR CARE® was used for nightly contact lens cleaning and disinfecting.
Period: Period 1, Approximately 30 Days
Arm/Group | LID210464, Then AOHG MF | AOHG MF, Then LID210464
Started | 51; 102 eyes | 50; 100 eyes
Completed | 50; 100 eyes | 50; 100 eyes
Not Completed | 1; 2 eyes | 0; 0 eyes
Not completed — Adverse Event | 1 | 0
Period: Period 2, Approximately 30 Days
Arm/Group | LID210464, Then AOHG MF | AOHG MF, Then LID210464
Started | 50; 100 eyes | 50; 100 eyes
Completed | 50; 100 eyes | 50; 100 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study according to actual study lens exposure.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID210464, Then AOHG MF | AOHG MF, Then LID210464 | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (6.9) | 50.0 (6.1) | 50.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 80
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 50 | 48 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 50 | 48 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Binocular High Contrast/High Illumination Visual Acuity at Distance With Study Lenses
Description: Visual acuity (VA) was assessed with study lenses in place under high contrast, high illumination. VA was collected for both eyes together using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 30, each wear period. A wear period was approximately 30 days.
Population: Full Analysis Set: All randomized subjects/eyes exposed to any study lenses evaluated in this study.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID210464: Lehfilcon A multifocal contact lenses (LID210464) worn in Period 1 or Period 2, as randomized, in both eyes for 30 days. CLEAR CARE® was used for nightly contact lens cleaning and disinfecting.
- AOHG MF: Lotrafilcon B multifocal contact lenses (AOHG MF) worn in Period 1 or Period 2, as randomized, in both eyes for 30 days. CLEAR CARE® was used for nightly contact lens cleaning and disinfecting.
Arm/Group | LID210464 | AOHG MF
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 100 | 100
logMAR | -0.10 (0.010) | -0.09 (0.010)
Statistical Analysis 1: Comparison: LID210464 vs AOHG MF; Test type: Non-Inferiority — Noninferiority in distance VA was declared if the least squares means difference upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least Squares Mean Difference = -0.01, 95% CI 1-sided [upper limit 0.00], Standard Error of Mean 0.006 — LSM results based on mixed effects repeated measures model with both fixed (lens, visit, lens-by-visit interaction, period, sequence, and habitual lens stratum) and random (subject) effects. Difference = LID210464 minus AOHG MF

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 60 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AE's is reported in units of eyes according to actual study lens exposure. All other populations are reported in units of subjects.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID210464 Ocular; LID210464 Non-Ocular: Events reported in this group occurred while exposed to the lehfilcon A contact lenses
- AOHG MF Ocular; AOHG MF Non-Ocular: Events reported in this group occurred while exposed to the lotrafilcon B contact lenses
Arm/Group | Pretreatment | LID210464 Ocular | LID210464 Non-Ocular | AOHG MF Ocular | AOHG MF Non-Ocular
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/202 | 0/101 | 0/200 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/202 | 0/101 | 0/200 | 1/100
Other Adverse Events (participants affected / at risk) | 0/101 | 0/202 | 0/101 | 0/200 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=101) | LID210464 Ocular (N=202) | LID210464 Non-Ocular (N=101) | AOHG MF Ocular (N=200) | AOHG MF Non-Ocular (N=100)
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT05338333/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT05338333/SAP_001.pdf